CLINICAL TRIAL: NCT07310355
Title: A Phase I/II, Single-Arm, Open-Label, Dose-Escalation and Expansion Study of 68Ga-PSMA-0057 and 177Lu-PSMA-0057 in Patients With PSMA-Positive Metastatic Castration-Resistant Prostate Cancer
Brief Title: 68Ga-PSMA-0057 and 177Lu-PSMA-0057 in Patients With PSMA-Positive Metastatic Castration-Resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu StarRay Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRT007-101
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA-0057 Treatment (Experimental): 1. Dose Escalation：Enroll patients with PSMA-positive progressive mCRPC who have received at least one novel endocrine therapy and 1-2 taxane-based treatment regimens, or are deemed intolerant by the investigator. Dose escalation will follow the "rolling six design" method, with two planned dose levels: 3.7 GBq and 6.0 GBq of fractionated 177Lu-PSMA-0057, administered every 6 weeks (Q6W), up to a maximum of 6 doses.
  2. Dose Expansion：After determining the RP2D of 177Lu-PSMA-0057, a phase II expansion will be conducted at the RP2D level (expected to expand only one dose level). Treatment will be administered every 6 weeks (Q6W), up to a maximum of 6 doses.
  Interventions: Drug: 68Ga-PSMA-0057; Drug: 177Lu-PSMA-0057

INTERVENTIONS:
Drug: 68Ga-PSMA-0057 — 68Ga-PSMA-0057 IV administered as imaging agent for PET/CT.
Drug: 177Lu-PSMA-0057 — 177Lu-PSMA-0057 radiopharmaceutical solution for injection.

SUMMARY:
This is a single-arm, open-label, Phase I/II clinical study designed to evaluate the safety, tolerability, pharmacokinetics, dosimetry, pharmacodynamics, and preliminary efficacy of Gallium [68Ga] PSMA-0057 Injection and Lutetium [177Lu] PSMA-0057 Injection as an integrated theranostic regimen in patients with PSMA-positive metastatic castration-resistant prostate cancer (mCRPC). The study consists of a Phase I dose-escalation phase to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of 177Lu-PSMA-0057, followed by a Phase II dose-expansion phase to further evaluate preliminary antitumor efficacy and confirm safety and pharmacologic profiles. Eligible participants will receive 68Ga-PSMA-0057 for PET imaging and 177Lu-PSMA-0057 for radioligand therapy. Key objectives include characterization of safety, tolerability, pharmacokinetics, dosimetry, pharmacodynamics, and preliminary therapeutic activity.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate well with investigators, understand the study purpose and requirements, voluntarily participate, and sign written informed consent.
2. Male, ≥18 years at screening.
3. Histologically or cytologically confirmed prostate cancer (excluding neuroendocrine prostate cancer and small cell prostate cancer), previously treated with at least one novel hormonal agent and 1-2 taxane-based regimens, or deemed intolerant to taxanes.
4. Serum/plasma testosterone at castrate level (<50 ng/dL or <1.7 nmol/L).
5. Documented progressive mCRPC based on ≥1 of the following: PSA progression (two consecutive PSA rises ≥1 week apart from a minimum value of 2.0 ng/mL); soft tissue progression per PCWG3 and RECIST v1.1; or bone progression with ≥2 new lesions.
6. PSMA-positive on imaging with 68Ga-PSMA-0057 (within 3 days before treatment start) or other investigator-accepted PSMA tracers (within 6 months before treatment start), using criteria in Section 4.8.5.
7. At least one measurable lesion per RECIST v1.1 and/or at least one bone metastasis per PCWG3.
8. Estimated life expectancy ≥12 weeks.
9. ECOG performance status 0-1 at baseline.
10. Adequate organ and bone marrow function, meeting the following lab criteria:

1)Bone Marrow: Absolute Neutrophil Count (ANC) ≥1.5×109/L, Platelets (PLT) ≥100×109/L, White Blood Cell (WBC) count ≥2.5×109/L, Hemoglobin (HGB) ≥9.0 g/dL (no transfusions/growth factors within 14 days prior to screening).

2)Liver Function: Serum Total Bilirubin (T-Bil) ≤1.5 ULN (unless Gilbert's syndrome); Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≤3 ULN for non-liver metastasis, or ≤5 ULN for liver metastasis.

3)Renal Function: Serum creatinine ≤1.5 ULN, or estimated Glomerular Filtration Rate (eGFR) ≥50 mL/min/1.73m2 (calculated using the MDRD formula).

11.Serum albumin concentration ≥30 g/L 12.Toxicities from prior therapies recovered to CTCAE v5.0 Grade 0-1 (alopecia excepted).

13.Men with reproductive potential agree to use highly effective contraception from informed consent through 6 months after last study dose and have no plans to donate sperm.

Exclusion Criteria:

1. History of hypersensitivity to any study drug component or excipients, or history of specific allergic disease requiring systemic therapy, or other serious allergic reactions.
2. Prior PSMA-targeted radioligand therapy, or treatment with radionuclides such as Sr-89, Sm-153, Re-186, Re-188, Ra-223, or hemibody radiation within 6 months prior to consent.
3. Use of any investigational drug or device within 30 days before consent.
4. Systemic anticancer therapy within 28 days or 5 half-lives prior to consent (whichever is longer), including chemotherapy, radiotherapy, immunotherapy, targeted therapy, systemic immunomodulatory drugs, or antitumor traditional Chinese medicines/formulations within 2 weeks before first dose.
5. Another malignancy within the past 5 years, except for curatively treated cervical carcinoma in situ, non-melanoma skin cancers, etc.
6. Major surgery or significant traumatic injury within 4 weeks before consent.
7. Active brain metastases or CNS involvement, including untreated symptomatic lesions or those requiring radiation, surgery, or steroids within 1 month prior to screening.
8. Symptomatic spinal cord compression or clinical/imaging findings suggestive of impending cord compression.
9. Severe arterial/venous thromboembolic events within 6 months prior to screening; history of stroke; uncontrolled hypertension; decompensated heart failure (NYHA III-IV); LVEF <50%; unstable angina; clinically significant arrhythmias requiring intervention.
10. Significant acute or chronic infections, including active TB, systemic bacterial or fungal infections requiring systemic therapy.
11. Clinically significant COPD or moderate-severe chronic respiratory disease requiring systemic therapy within 6 months before first dose.
12. Uncontrolled bladder outlet obstruction or incontinence (patients managed effectively with standard measures are allowed).
13. Active autoimmune disease requiring systemic treatment within the past 2 years or likely to recur, or active peptic ulcer disease or bleeding disorders.
14. History of solid organ transplantation or allogeneic hematopoietic stem cell transplantation (corneal transplant recipients not requiring immunosuppressants may be included).
15. Syphilis, HIV infection, HCV (HCV antibody positive with detectable HCV RNA), or active HBV infection (HBsAg positive with HBV DNA ≥ULN).
16. Contraindications to PET-CT or SPECT-CT imaging, or factors deemed by the investigator to preclude adequate imaging acquisition and interpretation.
17. Any condition judged by the investigator likely to interfere with compliance or study participation, or impair the ability to give informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 49 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events [68Ga-PSMA-0057] | 3 days
  Number of participants with adverse events as assessed by NCI-CTCAE v5.0
Incidence of adverse events [177Lu-PSMA-0057] | up to 2 years
  Number of participants with adverse events as assessed by NCI-CTCAE v5.0
Incidence of dose limiting toxicities [177Lu-PSMA-0057] | 6 weeks
  Number of participants with dose limiting toxicities
Preliminary efficacy: PSA50 response rate (Phase II) | up to 2 years
  Proportion of patients achieving ≥50% reduction in prostate-specific antigen (PSA) from baseline.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (demographics, safety, PK/PD, efficacy) will be shared upon reasonable request after publication of the primary results. Access requires a signed Data Use Agreement and sponsor approval. Requests should be submitted to clinicaltrials@starray.com
Time Frame: Data will be available starting 6 months after publication of primary results and for up to 5 years.